CLINICAL TRIAL: NCT01788527
Title: Continuous Glucose Monitoring in Women With Type 1 Diabetes in Pregnancy Trial
Acronym: CONCEPTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Sunnybrook Research Institute (Other); Jaeb Center for Health Research (Other); Cambridge University Hospitals NHS Foundation Trust (Other); University of Cambridge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-0037-A; NCT01734031 (obsolete NCT alias)
Record Dates: First submitted 2012-12-19; First posted 2013-02-11 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Type 1 Diabetics Who Are Pregnant or Planning Pregnancy
Keywords: Diabetes; Type 1; CGM; Continuous Glucose Monitor; HGM; HbA1c
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CGM (Experimental): Continuous Glucose Monitoring
  Interventions: Device: CGM
- HGM (No Intervention): Standard of care, Home Glucose Monitoring

INTERVENTIONS:
Device: CGM — Real Time Continuous Glucose Monitoring
  Arms: CGM

SUMMARY:
The primary objective of the study is to determine if RT CGM (Real Time-Continuous Glucose Monitoring) can improve glycemic control in women with T1D who are pregnant or planning pregnancy.

DETAILED DESCRIPTION:
In women with diabetes, hyperglycemia is associated with increased rates of numerous maternal and fetal adverse outcomes. Mothers are at increased risk of preeclampsia, polyhydramnios, and caesarean sections. Infants of mothers with diabetes have increased rates of congenital anomalies, premature delivery, macrosomia, stillbirth and NICU admissions. Macrosomia itself is associated with numerous adverse fetal outcomes including shoulder dystocia, birth injury, neonatal hypoglycemia, hyperbilirubinemia, respiratory distress syndrome and NICU admissions, asphyxia and death. Postprandial blood sugars in particular have been associated with increased macrosomia rates.

Numerous studies have shown that pregnancy outcomes can be reduced with improved glycemic control. In particular, pre-pregnancy care has been shown to assist women improve glucose control during the crucial period of organogenesis, and is associated with reduced rates of adverse pregnancy outcome including major congenital malformation, stillbirth and neonatal death.

Technological advances aimed at reducing glycemic excursions and improving glucose control in patients with diabetes include the continuous glucose monitoring (CGM) system. We hypothesize that real-time CGM will assist women with type 1 diabetes to improve their glycemic control before and during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes and using daily insulin therapy for at least one year
* Age 18-40 years
* Insulin regimen involves either the use of an insulin pump or multiple daily injections of insulin (at least 3 shots per day). Subjects using premixed fixed doses of insulin at the time of enrolment will not be eligible. Insulin regimen must be stable for at least 4 weeks (i.e. on multiple insulin injections or on insulin pump) prior to randomization.
* No expectation that subject will be moving out of the area of the clinical center during the next year, unless the move will be to an area served by another study center
* Informed Consent Form signed by the subject

In addition, specific eligibility criteria apply to the respective groups:

Pre-pregnancy Group:

* Patients who are planning pregnancy and wish to optimise glycemic control before conception

Pregnancy Group:

* Pregnancy gestation ≤13 weeks, 6 days at time of randomization
* Live singleton fetus
* Dating ultrasound (US) done to confirm gestational age, viability and rule out multiples. Gestational age will be based on the last menstrual period (LMP) provided there is a ≤5 day discrepancy with US dates in the first trimester and ≤10 day discrepancy with US dates in the second trimester. If the dates from LMP are outside these limits, the US dates will be used as the best estimate of gestational age.

Exclusion Criteria:

* Type 2 diabetes
* Gestational diabetes
* Previous participation in the study
* Estimated GFR <60 ml/min/1.73
* The presence of a significant medical disorder or use of a medication such as oral glucocorticoids that in the judgment of the investigator will affect the wearing of the sensors or the completion of any aspect of the protocol.

If the investigator is uncertain whether the patient would be eligible; i.e. if the medical disorder would constitute an exclusion, the Steering Committee will be asked to make the decision.

* Inpatient psychiatric treatment in the past 6 months
* Subjects using premixed fixed doses of insulin at the time of enrolment

In addition, specific exclusion criteria apply to the respective groups:

Pre-pregnancy Group:

* HbA1c <7.0% or >10.0%

Pregnancy Group:

* HbA1c <6.5% or >10.0%
* Known current higher order pregnancies (twins, triplets, etc.) These women will be excluded as they have a higher rate of adverse outcomes and could lead to inequalities if they are unequally distributed between the groups.
* Known potentially major fetal anomaly (as per EUROCAT criteria).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 325 (Actual)
Dates: Start 2013-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Glycemic Control in pre-pregnant group | 24 weeks or at conception
  Glycemic control as measured by HbA1c at 24 weeks or at conception. If the patient becomes pregnant, than a HbA1c will be measured post-confirmation of a positive pregnancy test and will contribute to the primary outcome.
Glycemic Control in pregnant group | 34 weeks gestation
  Glycemic control as measured by HbA1c at 34 weeks gestation. In women who do not progress to 34 weeks gestation, the latest measured HbA1c will be used to contribute to the primary outcome.

SECONDARY OUTCOMES:
Time in target in pre-pregnant group | 12 and 24 weeks after randomization
  Time in target at 12 and 24 weeks after randomization
HbA1c and time in target, in pre-pregnant group who became pregnant within 24 weeks from randomization | 24 weeks and 34 weeks gestation
  HbA1c and Time in target at post-confirmation of a positive pregnancy test, 24 weeks and 34 weeks gestation for those who start pre-pregnant and become pregnant
Time in target in pregnant group | Randomization, 24 weeks and 34 weeks gestation
  Time in target at randomization, 24 weeks and 34 weeks gestation
HbA1c measurement in pregnant group | 24 weeks and 34 weeks gestation
  HbA1c at randomization, 24 weeks and 34 weeks gestation
Hypertension in pregnant group | Up to 42 weeks gestation
  Incidence of worsening chronic hypertension, gestational hypertension, preeclampsia; total and individual measures
Caesarean sections in pregnant group | At delivery
  Caesarean section: primary and total
Gestational weight gain in pregnant group | Up to 34 weeks gestation
  Entry to 34 weeks gestation; 16 weeks to 34 weeks gestation
AUC | At delivery
  Area under the curve for blood sugars (a) >7.8 mmol/l or 140 mg/dl (b)>6.7 mmol/l or 120 mg/dl (c) <3.5 mmol/L or <63 mg/dl (d) <2.8 mmol/L or <50 mg/dl
Incidence of Clinical events | Up to 42 weeks gestation
  Episodes of 'severe hypoglycemia' requiring assistance; mild-moderate episodes of hypoglycemia <3.5 (mild) and <2.8 (moderate) from CGM data defined as AUC <3.5 or AUC less than or equal to 2.8 for 20 minutes duration; nocturnal hypoglycemia (NH) defined as CGM glucose <3.5 (mild) and <2.8 (moderate) between the hours of 23.00-07.00
Glucose variability | Up to delivery
  Mean amplitude of glycemic excursions (MAGE); Coefficient of Variation (CV); Standard deviation (SD) of CGM measurements; mean absolute rate of change of CGM based on one week of sensor values
Hospital stay | Admission until hospital discharge
  Length of hospital stay
Infant Outcomes | At birth of infant
  Infant birthweight >90th centile using customized growth curves; infant birthweight <10th centile using customized growth curves; infant birthweight >=4kg
Infant Outcomes | =<28 days of life
  Pregnancy loss (Miscarriage, stillbirth, neonatal death)
Infant Outcomes | At birth
  Preterm delivery (<37 weeks and early preterm <34 weeks)
Infant Outcomes | Until hospital discharge
  Birth injury
Infant outcomes | Until hospital discharge
  Shoulder dystocia
Infant outcomes | Until hospital discharge
  Neonatal hypoglycemia with intravenous dextrose
Infant Outcomes | Within first 7 days of life
  Hyperbilirubinemia
Infant Outcomes | Within first 7 days of life
  Respiratory Distress Syndrome (RDS)
Infant Outcomes | Until hospital discharge
  NICU admission > 24 hrs
Infant Outcomes | At birth
  Cord blood gas pH <7.0
Infant Outcomes | At birth
  Hyperinsulinemia (using Cord C-peptide)
Infant Outcomes | Within first 7 days of life or until hospital discharge (whichever is last)
  Composite fetal outcome: pregnancy loss:miscarriage, stillbirth, neonatal death (death<=28 days of life), birth injury, neonatal hypoglycemia, hyperbilirubinemia, respiratory distress syndrome requiring therapy, NICU admission >24 hours
Infant Outcomes | Within first 3 days of life
  Sum of skinfolds >90th percentile for gestational age
Infant Outcomes | Within first 3 days of life
  Other anthropometric measures
Infant Outcomes | Until hospital discharge
  Length of hospital stay
Insulin requirements | Pre-pregnant (randomization, 12 weeks, 24 weeks); Pregnant (randomization, 24 weeks and 34 weeks gestation)
  Units per kg per day
Questionnaires | Baseline and 24 weeks or at confirmed pregnancy (pre-pregnant); Baseline and 34 weeks (pregnant)
  BGMSRQ, HFS, PAID, SF12, CGM-SAT; NWTSQ
Study Contacts | Up to delivery
  Scheduled and unscheduled visits

CONTACTS AND LOCATIONS:
Overall Officials: Denice Feig, MD, Principal Investigator — MOUNT SINAI HOSPITAL; Helen Murphy, MB BCh BAO FRACP MD, Principal Investigator — Cambridge University Hospital NHS Foundation Trust and University of Cambridge
Locations (31):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States
- Canada (11):
  - Alberta Health Services - Calgary Zone, Calgary, Alberta
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster University, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - St Joseph's Health Care, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - St-Luc Hospital- Centre hospitalier de L'Universite de Montreal, Montreal, Quebec
  - Chuq-Chul, Québec, Quebec
  - Royal University Saskatoon, Saskatoon, Saskatchewan
- Galway University Hospital, Galway, Ireland
- Niguarda Ca' Granda Hospital, Milan, Italy
- Hospital De La Santa Creu I Sant Pau, Barcelona, Spain
- United Kingdom (16):
  - University of Aberdeen, Aberdeen, Scotland
  - Royal Infirmary of Edinburgh, Edinburgh, Scotland
  - Glasgow Royal Infirmary, Glasgow, Scotland
  - Russells Hall Hospital, Dudley, West Midlands
  - Addenbrooke's Hospital, Cambridge
  - Ipswich Hospital NHS Trust, Ipswich
  - St James University Hospital, Leeds
  - Guys & St. Thomas', London
  - Kings College Hospital, London
  - Manchester University Hospital NHS Trust, Manchester
  - South Tees Hospital NHS Trust, Middlesbrough
  - Royal Victoria Infirmary, Newcastle
  - Norfolk and Norwich University Hospital, Norwich
  - Queen's Medical Centre, Nottingham
  - Sheffield Teaching Hospitals, Sheffield
  - Princess Anne Hospital, Southampton

REFERENCES:
- [Derived] Ahmed RJ, Gafni A, Hutton EK, Hu ZJ, Sanchez JJ, Murphy HR, Feig DS; CONCEPTT Collaborative Group. The cost implications of continuous glucose monitoring in pregnant women with type 1 diabetes in 3 Canadian provinces: a posthoc cost analysis of the CONCEPTT trial. CMAJ Open. 2021 Jun 4;9(2):E627-E634. doi: 10.9778/cmajo.20200128. Print 2021 Apr-Jun. PMID 34088734
- [Derived] Tundidor D, Meek CL, Yamamoto J, Martinez-Bru C, Gich I, Feig DS, Murphy HR, Corcoy R; CONCEPTT Collaborative Group. Continuous Glucose Monitoring Time-in-Range and HbA1c Targets in Pregnant Women with Type 1 Diabetes. Diabetes Technol Ther. 2021 Oct;23(10):710-714. doi: 10.1089/dia.2021.0073. Epub 2021 May 25. PMID 33945304
- [Derived] Meek CL, Corcoy R, Asztalos E, Kusinski LC, Lopez E, Feig DS, Murphy HR; CONCEPTT collaborative group. Which growth standards should be used to identify large- and small-for-gestational age infants of mothers with type 1 diabetes? A pre-specified analysis of the CONCEPTT trial. BMC Pregnancy Childbirth. 2021 Jan 29;21(1):96. doi: 10.1186/s12884-021-03554-6. PMID 33514342
- [Derived] Meek CL, Tundidor D, Feig DS, Yamamoto JM, Scott EM, Ma DD, Halperin JA, Murphy HR, Corcoy R; CONCEPTT Collaborative Group. Novel Biochemical Markers of Glycemia to Predict Pregnancy Outcomes in Women With Type 1 Diabetes. Diabetes Care. 2021 Mar;44(3):681-689. doi: 10.2337/dc20-2360. Epub 2021 Jan 25. PMID 33495292
- [Derived] Neoh SL, Yamamoto JM, Feig DS, Murphy HR; CONCEPTT Collaborative Group. Dietary Patterns of Insulin Pump and Multiple Daily Injection Users During Type 1 Diabetes Pregnancy. Diabetes Care. 2020 Jan;43(1):e5-e7. doi: 10.2337/dc19-1908. Epub 2019 Nov 6. No abstract available. PMID 31694860
- [Derived] Feig DS, Donovan LE, Corcoy R, Murphy KE, Amiel SA, Hunt KF, Asztalos E, Barrett JFR, Sanchez JJ, de Leiva A, Hod M, Jovanovic L, Keely E, McManus R, Hutton EK, Meek CL, Stewart ZA, Wysocki T, O'Brien R, Ruedy K, Kollman C, Tomlinson G, Murphy HR; CONCEPTT Collaborative Group. Continuous glucose monitoring in pregnant women with type 1 diabetes (CONCEPTT): a multicentre international randomised controlled trial. Lancet. 2017 Nov 25;390(10110):2347-2359. doi: 10.1016/S0140-6736(17)32400-5. Epub 2017 Sep 15. PMID 28923465
- [Derived] Feig DS, Asztalos E, Corcoy R, De Leiva A, Donovan L, Hod M, Jovanovic L, Keely E, Kollman C, McManus R, Murphy K, Ruedy K, Sanchez JJ, Tomlinson G, Murphy HR; CONCEPTT Collaborative Group. CONCEPTT: Continuous Glucose Monitoring in Women with Type 1 Diabetes in Pregnancy Trial: A multi-center, multi-national, randomized controlled trial - Study protocol. BMC Pregnancy Childbirth. 2016 Jul 18;16(1):167. doi: 10.1186/s12884-016-0961-5. PMID 27430714